CLINICAL TRIAL: NCT05953480
Title: A Phase 2b, Multinational, Randomized, Double-blind Study to Investigate the Efficacy and Safety of Redasemtide (S-005151) Compared With Placebo in Adult Participants With Acute Ischemic Stroke
Brief Title: A Phase 2b, Randomized, Double-blind Study of Redasemtide (S-005151) in Adult Participants With Acute Ischemic Stroke
Acronym: Revive
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2138P2231; 2022-501890-38-00 (Registry Identifier: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Redasemtide; S-005151; Plasminogen activator; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Redasemtide Dose A (Experimental): Redasemtide will be administered as an intravenous (IV) infusion once daily for 5 consecutive days during hospitalization.
  Interventions: Biological: Redasemtide
- Redasemtide Dose B (Experimental): Redasemtide will be administered as an IV infusion once daily for 5 consecutive days during hospitalization.
  Interventions: Biological: Redasemtide
- Placebo (Placebo Comparator): Placebo will be administered in an amount equivalent to redasemtide, as an IV infusion, once daily for 5 consecutive days during hospitalization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Redasemtide — Lyophilized white powder reconstituted in 0.9% saline for injection
  Other Names: Redasemtide trifluoroacetate; S-005151
  Arms: Redasemtide Dose A; Redasemtide Dose B
Drug: Placebo — Lyophilized white powder reconstituted in 0.9% saline for injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of redasemtide in adult participants with acute ischemic stroke (AIS). This study consists of 2 cohorts, Cohort A and Cohort B. Cohort A (redasemtide or placebo) will enroll participants who are ineligible for systemic thrombolysis and/or mechanical recanalization therapy. Cohort B (redasemtide or placebo) will enroll participants who are eligible to receive or who have received systemic thrombolysis and/or mechanical recanalization therapy as standard of care.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to initiate study intervention within 25 hours of stroke onset
* Cohort A: Determined by the investigator to not be eligible for systemic thrombolysis and/or mechanical recanalization therapy (that is, mechanical thrombectomy, local fibrinolytic therapy as per local standard of care) for the current stroke.
* Cohort B: Determined by the investigator to be eligible for systemic thrombolysis and/or mechanical recanalization therapy (that is, mechanical thrombectomy, local fibrinolytic therapy as per local standard of care) for the current stroke.
* Cohort A: If a participant is not eligible for systemic thrombolysis and/or mechanical recanalization therapy, screening and baseline NIHSS score of 6 to 22 is required (inclusive) and must be stable, defined as absence of an increase or decrease of ≥4 points within ≥1 hour to ≤3 hours of screening, and NIHSS score should be 6 to 22 at baseline.
* Cohort B: In a participant who is eligible to receive or has received concomitant systemic thrombolysis and/or mechanical recanalization therapy, the NIHSS score must be 6 to 22 at screening prior to systemic thrombolysis and/or mechanical recanalization therapy and the second/baseline NIHSS score must be 6 to 22 and should be done after systemic thrombolysis and/or mechanical recanalization therapy.
* Medically stable at the time of enrollment except for primary disease and complications associated with it, according to the judgment of the investigator. In addition, hospitalization during the Follow-up Period is not anticipated, and the participant appears likely to be able to complete the study. Medically stable is defined as disease not requiring significant change in therapy for 3 months following enrollment.

Key Exclusion Criteria:

* Any disease or neurological disorder that, in the opinion of the investigator, would interfere with the conduct of the study
* A severe decrease in consciousness level (defined as NIHSS item 1a score 3: Not alert, responds only with reflex motor or autonomic effects, or totally unresponsive, flaccid, and areflexic)
* Disability corresponding to a mRS score of ≥2 before the onset of stroke
* A history of stroke (excluding transient ischemic attack), history of or current intracranial hemorrhage, or head trauma that caused neurological effects within 90 days prior to obtaining informed consent
* Participants with an ischemic stroke in cerebellum and/or brain stem as the main infarction site
* Diagnosis of a current transient ischemic attack
* Unable to undergo either computed tomography or magnetic resonance imaging
* Considered by the investigator to be inappropriate to participate due to a history or complication of serious cardiovascular disease within 1 month of screening (for example, history of acute myocardial infarction, current acute myocardial infarction, uncontrollable heart failure, infective endocarditis requiring treatment, or acute aortic dissection, or requiring or likely to require hospitalization for severe arrhythmia during the study)
* Blood glucose level <50 or >400 milligrams/deciliter after glycemic control
* Systolic blood pressure ≥220 millimeters of mercury (mmHg) or diastolic blood pressure ≥120 mmHg after antihypertensive treatment
* Sensitivity to any of the study interventions, or components thereof, or clinically significant drug or other severe allergy that, in the opinion of the investigator, contraindicates participation in the study
* Use of prohibited concomitant medications or therapies listed in the protocol for the treatment of current AIS
* Participants who have previously received redasemtide
* Participants who have received any investigational product within 90 days of screening

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) Score at Day 90 | Day 90

SECONDARY OUTCOMES:
Number of Participants With mRS Score of 0 to 2 | Day 90
Number of Participants With Barthel Index (BI) Score ≥ 95 | Day 90
mRS Score at Day 30 | Day 30
mRS Score at Day 180 | Day 180
Number of Participants With National Institutes of Health Stroke Scale (NIHSS) Score of 0 or 1 | Days 1, 5, 30, 90, and 180
Change From Baseline in NIHSS Score | Baseline, Days 1, 5, 30, 90, and 180
Number of Participants With BI Score ≥ 95 | Days 5, 30, and 180
Change From Day 5 in Short Form 36-item Health Survey (SF-36) Score | Day 5, Days 90 and 180
Change From Day 5 in Stroke and Aphasia Quality of Life Scale - 39 Item Generic Version (SAQoL-39g) Score | Day 5, Days 90 and 180
Patient Global Impression of Change Scale (PGI-C) Score | Days 5, 90, and 180
Change From Day 5 in Patient Global Impression of Severity Scale (PGI-S) Score | Day 5, Days 90 and 180

CONTACTS AND LOCATIONS:
Locations (150):
- United States (17):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Intercoastal Medical Group, Sarasota, Florida
  - Augusta University, Augusta, Georgia
  - Mercyhealth Javon Bea Hospital- Riverside, Rockford, Illinois
  - Community Hospital, Munster, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Munson Healthcare, Traverse City, Michigan
  - Mayo Clinic Hospital-Rochester, St. Mary's Campus - PPDS, Rochester, Minnesota
  - North Shore University Hospital-300 Community Dr, Manhasset, New York
  - Nuvance Health Medical Practice, PC- Neurosurgery, Poughkeepsie, New York
  - Summa Health System - Akron Campus, Akron, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Baylor University Medical Center - 3500 Gaston Ave, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Scott & White - Plano Brain & Spine Center, Plano, Texas
  - University Health-University Hospital, San Antonio, Texas
- Australia (6):
  - Liverpool Hospital - PPDS, Sydney, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - UZ Brussel - PIN, Jette, Brussels Capital
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Oostende - Damiaan, Ostend, West-Vlaanderen
- China (6):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
- Czechia (3):
  - Vseobecna Fakultni Nemocnice V Praze-U Nemocnice 499/2, Prague, Nové Město
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha, Hlavní Mesto
  - Fakultni nemocnice v Motole, Prague
- Helsingin yliopistollinen sairaala, Helsinki, Uusimaa, Finland
- Germany (2):
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
- Greece (12):
  - University General Hospital of Patras, Pátrai, Achaïa
  - Naval Hospital of Athens, Athens, Attica
  - Alexandra Hospital, Athens, Attica
  - University General Hospital of Alexandroupolis, Alexandroupoli, Evros
  - University General Hospital of Heraklion, Heraklion, Irakleio
  - University General Hospital ''ATTIKON'', Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki ''Hippokratio'', Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki ''G. Papanikolaou'', Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital - PPDS, Hong Kong
  - Princess Margaret Hospital - Hong Kong, Kwai Chung
  - Prince of Wales Hospital, Shatin
- Hungary (8):
  - Pécsi Tudomanyegyetem - Vasvari Pal u., Pécs, Baranya
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz és Egyetemi Oktatokorhaz, Miskolc, Borsod-Abauj Zemplen county
  - Kistarcsai Flór Ferenc Kórház, Kistarcsa, Pest County
  - Szent Damjan Gorogkatolikus Korhaz, Kisvárda, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem, Budapest
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Semmelweis Egyetem Idegsebeszeti es Neurointervencios Klinika, Budapest
  - Gyor-Moson-Sopron Varmegyei Petz Aladár Egyetemi Oktató Kórház, Győr
- Israel (9):
  - Meir Medical Center, Kfar Saba, Central District
  - Hillel Yaffe Medical Center, Hadera, Haifa District
  - Hadassah Medical Center - PPDS, Jerusalem, Jerusalem
  - Galilee Medical Center, Nahariya, Northern District
  - Tel Aviv Sourasky Medical Center - PPDS, Tel Aviv, Tel Aviv
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center - PPDS, Haifa
  - Sheba Medical Center - PPDS, Ramat Gan
  - ZIV Medical Center, Safed
- Japan (27):
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Social Medical Corporation The Chiyukai Foundation Fukuoka Wajiro Hospital, Fukuoka, Fukuoka
  - Shin Komonji Hospital, Kitakyushu-Shi, Fukuoka
  - Omuta City Hospital, Omuta-Shi, Fukuoka
  - Japanese Red Cross Takayama Hospital, Takayama-Shi, Gifu
  - National Hospital Organization Higashihiroshima Medical Center, Higashihiroshima-Shi, Hiroshima
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure-Shi, Hiroshima
  - Fukui Prefectural Hospital, Fukui-shi, Hukui
  - Our Lady of the Snow Social Medical Corporation St. Mary's Hospital, Kurume-Shi, Hukuoka
  - Shinsuma General Hospital, Kobe, Hyôgo
  - Hyogo Medical University Hospital, Nishinomiya-Shi, Hyôgo
  - Seisho Hospital, Odawara-Shi, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - National Hospital Organization Beppu Medical Center, Beppu-Shi, Oita Prefecture
  - Rinku General Medical Center, Izumisano, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - Tominaga Hospital, Osaka, Osaka
  - National Cerebral and Cardiovascular Center, Suita-Shi, Osaka
  - Osaka University Hospital, Suita-Shi, Osaka
  - Shin-Kuki General Hospital, Kuki-shi, Saitama
  - National Hospital Organization Hamada Medical Center, Hamada-Shi, Shimane
  - Shizuoka City Shizuoka Hospital, Aoi-Ku, Shizuoka
  - Japan Organization of Occupational Health and Safety Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - Chutoen General Medical Center, Kakegawa-Shi, Shizuoka
  - Misyuku Hospital, Meguro-Ku, Tokyo
  - Sanyudo Hospital, Yonezawa-Shi, Yamagata
- Serbia (11):
  - Hospital for Cerebrovascular Diseases Sveti Sava, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia - Pasterova 2 - PPDS, Belgrade
  - General Hospital Bor, Bor
  - General Hospital Cuprija, Ćuprija
  - General Hospital Leskovac, Leskovac
  - University Clinical Center Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad
  - Health Center Uzice, Užice
  - Health Center Valjevo, Valjevo
  - General Hospital Dr. Djordje Joanovic - Zrenjanin, Zrenjanin
- Singapore (2):
  - National University Hospital- Singapore, Singapore
  - Singapore General Hospital (SGH), Singapore
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu, Daegu Gwang'yeogsi
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggido
  - Pusan National University Hospital, Busan
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Hanyang University Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (22):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Torrecardenas, Almería
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (11):
  - Aberdeen Royal Infirmary - PPDS, Aberdeen, Aberdeenshire
  - Luton and Dunstable Hospital, Luton, Bedfordshire
  - Royal Berkshire Hospital NHS Foundation Trust, Reading, Berkshire
  - Charing Cross Hospital, London, London, City of
  - Northwick Park Hospital, Harrow, Middlesex
  - The Royal London Hospital, London, Middlesex
  - National Hospital for Neurology & Neurosurgery, London, Middlesex
  - King's College Hospital, London, Surrey
  - Fairfield General Hospital - PPDS, Bury
  - Leicester Royal Infirmary, Leicester
  - Royal Victoria Infirmary, Newcastle

IPD SHARING:
Plan to Share IPD: No